CLINICAL TRIAL: NCT05845931
Title: Sex Differences in Berberine Pharmacokinetics in Healthy Volunteers - BERKI-2
Brief Title: Sex Differences in Berberine Pharmacokinetics
Acronym: BERKI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Stefan Engeli, MD, Prof. Dr. med Stefan Engeli, University Medicine Greifswald
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPHA-2023-006
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetic Study in Healthy Volunteers
Keywords: Berberine; Sex differences; pharmacokinetic; menstrual cycle
MeSH Terms: interventions — Berberine

STUDY DESIGN:
Intervention Model Description: This is an unblinded, non-randomized, prospective Kinetic study comparing age-matched women and men (parallel). In women, an additional cross-over approach is applied
Masking Description: This Study will be an open label study. Participants will be selected from an existing database of our Institute.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- woman (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between arm 1 and arm 2.
  Interventions: Dietary Supplement: Berberine
- men (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between arm 1 and arm 2.
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Dietary Supplement: Berberine — A single dose of 1000 mg berberine in two capsules will be administered with 250 ml of still water in the overnight fasting condition. A total of 11 blood samples will be taken at defined time points (baseline, 1; 1.5; 2; 3; 4; 5; 6; 8; 10; 24 h). At each time point, blood will be collected in 2x 7.5 ml tubes for collecting serum and plasma samples to determine berberine concentrations. (Women will undergo the Intervention twice, once in the 1st half and once in the 2nd half of their menstrual cycle.) In addition urine will be collected over the time of 0-10 h after berberine intake and body composition will be measured by bioelectrical impedance analysis (BIA).

SUMMARY:
The influence of genetic variants of the CYP2D6 enzyme and the Organic Cation Transporter 1 on the kinetics of berberine (BERKI-1) has recently been studied. By chance, a significant sex difference was observed independent of the genetic variant. The Area under the curve of berberine in women compared to men was about three times higher, and the difference was statistically significant

The aim of BERKI-2 is to confirm the sex difference in an independent second study. In addition, influences of sex hormones on berberine kinetics in women will be studied.

As in BERKI-1, time-dependent blood and urine samples will be collected after a single berberine dose. By measuring berberine metabolites by Liquid Chromatography and Mass-spectrometry standard kinetic parameters e.g., AUC0-24, Cmax, Tmax will be calculated. Age-matched healthy women (n = 15) and men (n = 15) will be enroled.

DETAILED DESCRIPTION:
A single dose of 1000 mg berberine will be administered in two capsules with 250 ml of still water in the overnight fasting condition at 8 a.m.. A total of 11 blood samples will be taken at defined time points (baseline, 1; 1.5; 2; 3; 4; 5; 6; 8; 10; 24; h). At each time point, blood will be collected in 2x 7.5 ml tubes for collecting serum and plasma samples to determine berberine concentrations. Another serum sample will be obtained at baseline from women only to determine estradiol, progesterone, luteinizing hormone and follicle stimulating hormone to characterize the first and second phase of the cycle.

Every hour, participants will drink 100 ml of sparkling water to stimulate intestinal peristalsis and promote transport of the capsule. Volunteers are asked to stay in bed during the first four hours but are then allowed to move freely within the Clinical Research Unit. After 2 h, participants may drink a cup of tea or coffee and after 4 h they will be served a meal. Urine will be collected during the first 10 h after administration. Between 2 and 4 p.m., measuring body composition by bioelectrical impedance analysis (BIA) will be peformed to obtain fat mass and fat free mass (total and percentage) and body water. We use the seca mBCA 525 scale.The participants will stay in the Clinical Research Unit of the Institute of Pharmacology for the first 10 h after administration.

Women will undergo this treatment twice at least one week apart. Once in the first half (between days 4-10 after start of menstrual bleeding) and once in the second half (between days 20-26 after start of menstrual bleeding) of their menstrual cycle. The first day of menstrual bleeding marks day 1 as a reference.

ELIGIBILITY:
Inclusion Criteria:

* wild type genotypes for CYP2D6 and Organic Cation Transporter 1
* understands the study purpose and design
* contractually capable and provides signed informed consent form
* healthy condition or mild and/or well treated forms of allergies, asthma, hypertension, and orthopaedic diseases
* no regular use of more than 2 drugs

Exclusion Criteria:

* volunteers who have already participated in BERKI-1
* BMI <18 kg/m2 and >35 kg/m2
* disorders of sex hormone regulation, hormone treatments
* women: menopause,known pregnancy or lactation period, positive urine pregnancy test at screening and at visits, oral contraceptives, depot contraceptives, or hormone-re-leasing intrauterine devices
* anaemia (haemoglobin < 13 g/dl (8,07 mmol/l) in men or < 12 g/dl (7,45 mmol/l) in women
* elevated liver function tests (> 2x ULN)
* reduced renal function (eGFRMDRD < 60 ml/min/1,7m2)
* psychiatric disease or drug dependency at time of visit
* use of recreational drugs more than twice a week
* poor venous conditions that make it impossible to place a peripheral venous catheter

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Berberine plasma concentration women vs. men | day 1
  Difference in berberine plasma concentrations expressed as Area under the Curve between women and men.

SECONDARY OUTCOMES:
Berberine plasma concentrations durig first and second half of the menstrual cycle | day 1
  Difference in berberine plasma concentrations expressed as Area under the Curve between the 1st and the 2nd phase of the female menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engeli, Prof., Principal Investigator — Universitätsmedizin Greifswald, Institut für Pharmakologie
Locations (1):
- Center of Drug Absorption and Transport (C_DAT), Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao Q, Wei T, Qiu H, Cai Y, Yuan L, Liu X, Li X. Epigenetic Effects of Natural Products in Inflammatory Diseases: Recent Findings. Phytother Res. 2025 Jan;39(1):90-137. doi: 10.1002/ptr.8364. Epub 2024 Nov 8. PMID 39513382